CLINICAL TRIAL: NCT00651430
Title: Step Execution, Stability, Quality of Life, Fear of Falling and Their Association Following Total Hip Arthroplasty
Brief Title: Physical Functioning Following Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Itshak Melzer PhD, PT, Ben-Gurion University of the Negev
Other Study IDs: sor462807ctil; MB4628
Record Dates: First submitted 2008-01-14; First posted 2008-04-02 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthrosis, Balance Control, Voluntary Movement Control
Keywords: Balance; Voluntary stepping; function; disability; fear of falls; Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no biospecimens are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A

SUMMARY:
Adults suffer from Osteoarthrosis of hip joint that willing to participate in the study will be tested with well-established measuring techniques of Balance control using force plate before 3 month and 6 month after Total Knee Arthroplasty (THA) in the movement and Rehabilitation Laboratory at BGU. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). Each of the Times (before 3 month and 6 month after the THA) in two task conditions (eyes closed and eyes close conditions). Participants will be required to stand on the platform 10 times for 30 s For each trial, they will be instructed to sway as little as possible. In addition step execution test and Late life function and disability questionnaires will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Able to stand safely for 30 seconds
* Able to walk independently
* Hip OA prior THA

Exclusion Criteria:

* Stroke or other neurological diseases
* Minimal score 24 or higher
* Blindness

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 adults suffer from Hip OA prior THA
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
SDF parameters | before, 3 month and 6 month after the THA

SECONDARY OUTCOMES:
Late Life Function and disability, Fall efficacy scale, step execution test | before 3 month and 6 month after

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Benkovich, MD, Study Director — Soroka University Medical Center; Itshak Melzer, PhD, PT, Principal Investigator — Ben-Gurion University of the Negev
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - SorokaUMC, Beersheba